CLINICAL TRIAL: NCT07353034
Title: Examining the Role of Functional Social Support Subtypes for Self-Management Capacity Among Individuals With COPD
Brief Title: Functional Social Support in COPD Self-Management
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00145926
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Social Support; Self-Management Capacity; Chronic Disease Management; Behavioral Health; Psychosocial Support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD Adults (≥40 years): Adults aged 40 years and older with a self-reported diagnosis or treatment for chronic obstructive pulmonary disease (COPD). All participants will complete an online survey; a subset will participate in qualitative interviews.

SUMMARY:
This observational study aims to examine how different types of functional social support (emotional/informational, tangible, affectionate, and positive social interaction) predict self-management capacity among individuals with chronic obstructive pulmonary disease (COPD). The study includes a quantitative cross-sectional survey and qualitative semi-structured interviews (N=20) to explore barriers and facilitators to adequate social support. Findings will inform the development of targeted self-management interventions for COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40
* Self-reported COPD diagnosis or treatment
* English-speaking
* Internet access

Exclusion Criteria:

* History of psychosis or severe mental illness
* Ongoing substance abuse
* Other chronic respiratory conditions (e.g., lung cancer, asthma)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 40 years and older with a self-reported diagnosis or treatment for chronic obstructive pulmonary disease (COPD). Participants must be English-speaking and have internet access to complete an online survey and, if selected, participate in a qualitative interview. Recruitment will occur through the Medical University of South Carolina health system and COPD Foundation online platforms.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-management capacity | At enrollment (single time point)
  Measured using the Chronic Respiratory Disease Questionnaire (CRQ) - Mastery domain; score range 1-7, where higher scores indicate greater perceived control over COPD symptoms.

SECONDARY OUTCOMES:
Functional social support subdomains | At enrollment
  Measured using Medical Outcomes Study Social Support Survey (MOS-SSS); subscale scores for emotional/informational, tangible, affectionate, and positive social interaction.
Structural social support | At enrollment
  Measured using Social Support Questionnaire - Short Form (SSQ-6).
Symptom severity | At enrollment
  Measured using COPD Assessment Test (CAT).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Morgan, BSN, RN, CEN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified aggregate data may be shared through publications and presentations; individual participant data will not be shared.